CLINICAL TRIAL: NCT01034995
Title: An Eight-week, Multinational, Multicenter, Double-blind, Active- and Placebo-controlled Clinical Trial Evaluating the Efficacy and Tolerability of Three Fixed Doses of SSR125543 (20 mg Daily, 50 mg Daily and 100 mg Daily) in Outpatients With Major Depressive Disorder
Brief Title: A Trial Evaluating the Efficacy and Tolerability of SSR125543 in Outpatients With Major Depressive Disorder
Acronym: AGATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DFI5687; 2009-010339-42 (Other: EMEA)
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — SSR125543; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- SSR125543 20 mg (Experimental): 1 capsule of SSR125543 20 mg + 1 capsule of placebo
  Interventions: Drug: SSR125543
- SSR125543 50 mg (Experimental): 1 capsule of SSR125543 50 mg + 1 capsule of placebo
  Interventions: Drug: SSR125543
- SSR125543 100 mg (Experimental): 2 capsules of SSR125543 50 mg
  Interventions: Drug: SSR125543
- escitalopram 10 mg (Active Comparator): 1 capsule of escitalopram 10 mg + 1 capsule of placebo
  Interventions: Drug: escitalopram
- placebo (Placebo Comparator): 2 capsules of placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SSR125543 — Pharmaceutical form: capsule
  Route of administration: oral
  Arms: SSR125543 100 mg; SSR125543 20 mg; SSR125543 50 mg
Drug: escitalopram — Pharmaceutical form: encapsulated tablets
  Route of administration: oral
  Arms: escitalopram 10 mg
Drug: placebo — Pharmaceutical form: capsule
  Route of administration: oral
  Arms: placebo

SUMMARY:
Primary Objective:

* To evaluate the efficacy of three fixed doses of SSR125543 (20 mg daily, 50 mg daily, and 100 mg daily) compared to placebo in outpatients with major depressive disorder, as assessed by the change from baseline (Day -1) to Day 56 in the 17-item Hamilton Depression Rating Scale (HAM-D) total score.

Secondary Objectives:

* To evaluate the tolerability and safety of SSR125543 in outpatients with major depressive disorder
* To evaluate plasma concentrations of SSR125543

DETAILED DESCRIPTION:
This duration of this trial is 11 weeks.

ELIGIBILITY:
Inclusion criteria:

* Patients with a diagnosis of major depressive disorder, as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR) criteria (296.3) and confirmed by the semi-structured Mini International Neuropsychiatric Interview (MINI).

Exclusion criteria:

* Inpatient hospitalization at screening
* Symptoms of depression present for <30 days or >2 years
* Significant suicide risk
* Mild depression as measured by standard clinical research scales
* History of failure to respond to antidepressant treatment
* Other psychiatric conditions that could obscure the results of the study
* For women of child-bearing potential, the unwillingness to use highly effective means of birth control

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 580 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline (Day -1) to Day 56 in the 17-item HAM-D total score | 8 weeks

SECONDARY OUTCOMES:
Change from baseline in HAM-D depressed mood item | 8 weeks
Change from baseline in HAM-D responders (50% improvement) | 8 weeks
Changes from baseline in the HAM-D core and factor scores | 8 weeks
Changes from baseline in the Montgomery-Asberg depression rating scale (MADRS) total score | 8 weeks
Changes from baseline in the Clinical Global Impression (CGI) Severity of Illness score | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (73):
- Belgium (3):
  - Sanofi-Aventis Investigational Site Number 056002, Asse
  - Sanofi-Aventis Investigational Site Number 056003, Brussels
  - Sanofi-Aventis Investigational Site Number 056001, Liège
- Canada (9):
  - Sanofi-Aventis Investigational Site Number 124011, Burlington
  - Sanofi-Aventis Investigational Site Number 124012, Chatham
  - Sanofi-Aventis Investigational Site Number 124004, Edmonton
  - Sanofi-Aventis Investigational Site Number 124003, Gatineau
  - Sanofi-Aventis Investigational Site Number 124001, Kelowna
  - Sanofi-Aventis Investigational Site Number 124006, Mississauga
  - Sanofi-Aventis Investigational Site Number 124008, Penticton
  - Sanofi-Aventis Investigational Site Number 124007, Sherbrooke
  - Sanofi-Aventis Investigational Site Number 124009, Toronto
- Chile (8):
  - Sanofi-Aventis Investigational Site Number 152001, Santiago
  - Sanofi-Aventis Investigational Site Number 152002, Santiago
  - Sanofi-Aventis Investigational Site Number 152003, Santiago
  - Sanofi-Aventis Investigational Site Number 152005, Santiago
  - Sanofi-Aventis Investigational Site Number 152006, Santiago
  - Sanofi-Aventis Investigational Site Number 152004, Santiago
  - Sanofi-Aventis Investigational Site Number 152007, Valparaíso
  - Sanofi-Aventis Investigational Site Number 152008, Viña del Mar
- Estonia (4):
  - Sanofi-Aventis Investigational Site Number 233001, Tallinn
  - Sanofi-Aventis Investigational Site Number 233002, Tallinn
  - Sanofi-Aventis Investigational Site Number 233004, Tallinn
  - Sanofi-Aventis Investigational Site Number 233003, Tartu
- Finland (5):
  - Sanofi-Aventis Investigational Site Number 246001, Helsinki
  - Sanofi-Aventis Investigational Site Number 246003, Helsinki
  - Sanofi-Aventis Investigational Site Number 246005, Jarvenpaa
  - Sanofi-Aventis Investigational Site Number 246002, Tampere
  - Sanofi-Aventis Investigational Site Number 246004, Turku
- France (8):
  - Sanofi-Aventis Investigational Site Number 250008, Arcachon
  - Sanofi-Aventis Investigational Site Number 250007, Dole
  - Sanofi-Aventis Investigational Site Number 250006, Élancourt
  - Sanofi-Aventis Investigational Site Number 250001, Grenoble
  - Sanofi-Aventis Investigational Site Number 250003, Montpellier
  - Sanofi-Aventis Investigational Site Number 250005, Nîmes
  - Sanofi-Aventis Investigational Site Number 250004, Orvault
  - Sanofi-Aventis Investigational Site Number 250002, Toulouse
- Germany (8):
  - Sanofi-Aventis Investigational Site Number 276008, Achim
  - Sanofi-Aventis Investigational Site Number 276002, Berlin
  - Sanofi-Aventis Investigational Site Number 276004, Dresden
  - Sanofi-Aventis Investigational Site Number 276005, Leipzig
  - Sanofi-Aventis Investigational Site Number 276006, Mannheim
  - Sanofi-Aventis Investigational Site Number 276007, München
  - Sanofi-Aventis Investigational Site Number 276001, Schwerin
  - Sanofi-Aventis Investigational Site Number 276003, Würzburg
- Sanofi-Aventis Investigational Site Number 528001, The Hague, Netherlands
- Russia (11):
  - Sanofi-Aventis Investigational Site Number 643006, Moscow
  - Sanofi-Aventis Investigational Site Number 643005, Nizhny Novgorod
  - Sanofi-Aventis Investigational Site Number 643008, Rostov-on-Don
  - Sanofi-Aventis Investigational Site Number 643001, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643009, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643010, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643011, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643003, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643002, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643004, Samara
  - Sanofi-Aventis Investigational Site Number 643007, Smolensk
- Slovakia (5):
  - Sanofi-Aventis Investigational Site Number 703102, Bratislava
  - Sanofi-Aventis Investigational Site Number 703101, Bratislava
  - Sanofi-Aventis Investigational Site Number 703104, Michalovce
  - Sanofi-Aventis Investigational Site Number 703105, Rimavská Sobota
  - Sanofi-Aventis Investigational Site Number 703103, Rožňava
- South Africa (6):
  - Sanofi-Aventis Investigational Site Number 710005, Cape Town
  - Sanofi-Aventis Investigational Site Number 710001, Cape Town
  - Sanofi-Aventis Investigational Site Number 710006, Centurion
  - Sanofi-Aventis Investigational Site Number 710002, Durban
  - Sanofi-Aventis Investigational Site Number 710003, Pretoria
  - Sanofi-Aventis Investigational Site Number 710004, Somerset West
- Sweden (5):
  - Sanofi-Aventis Investigational Site Number 752004, Linköping
  - Sanofi-Aventis Investigational Site Number 752002, Lund
  - Sanofi-Aventis Investigational Site Number 752003, Malmo
  - Sanofi-Aventis Investigational Site Number 752005, Stockholm
  - Sanofi-Aventis Investigational Site Number 752001, Uppsala